CLINICAL TRIAL: NCT07178249
Title: A Phase I/II Clinical Study Evaluating the Safety and Preliminary Efficacy of EXG202 in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: Evaluating the Safety and Preliminary Efficacy of EXG202 Gene Therapy for Neovascular AMD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hangzhou Jiayin Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EXG202-111
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Wet Age-related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose escalation-Cohort 1 (Experimental): Dose 1 :Administered via intravitreal injection
  Interventions: Biological: EXG202 injection
- Dose escalation-Cohort 2 (Experimental): Dose 2 :Administered via intravitreal injection
  Interventions: Biological: EXG202 injection
- Dose escalation-Cohort 3 (Experimental): Dose 3 :Administered via intravitreal injection
  Interventions: Biological: EXG202 injection
- Dose escalation-Cohort 4 (Experimental): Dose 4 :Administered via intravitreal injection
  Interventions: Biological: EXG202 injection

INTERVENTIONS:
Biological: EXG202 injection — EXG202 injection is a gene therapy product for the treatment of wet (neovascular) Age-related Macular Degeneration（wAMD） with a single intravitreal injection and administration.

SUMMARY:
VEGF inhibitors (anti-VEGF),such as aflibercept has been shown to be safe and effective for treating nAMD and have demonstrated improvement in vision. However, anti-VEGF therapy is administered frequently via intravitreal injection and can be a significant burden to the patients.

EXG 202 is a recombinant adeno-associated virus (rAAV) gene therapy vector carrying a coding sequence for a soluble anti-VEGF protein. The long-term, stable delivery of this therapeutic protein following a 1 time gene therapy treatment for nAMD could potentially reduce the treatment burden of currently available therapies while maintaining vision with a favorable benefit.

DETAILED DESCRIPTION:
This Phase I/II study was designed to evaluate the safety and Preliminary Efficacy of EXG202 gene therapy in subjects with nAMD. Subjects who met the inclusion/exclusion criteria and had response to an initial anti-VEGF injection received a single dose of EXG202 administered . Safety was the primary focus for the phase I/II trial ,at the same time ,preliminary Efficacy also is another goal for the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥50 years old;
2. The study eye must be diagnosed of wAMD and current active lesions;
3. Subjects have clear refractive media and sufficient pupil dilation at the time of screening to obtain high-quality retinal images for confirmation of diagnosis;
4. Subjects (including male subjects) have no pregnancy plans during the screening period and the entire trial period and voluntarily take effective contraceptive measures and have no sperm or egg donation plans;
5. Subjects are Voluntarily participate in this clinical trial, understand the research procedures and sign the informed consent form before screening; subjects have good compliance and are willing to abide by the research procedures.

Exclusion Criteria:

1. The study eye has any eye disease other than wAMD that may affect central vision and/or macular detection ;
2. The study eye has a history of retinal detachment or retinal detachment during the screening period;
3. The study eye has MNV caused by reasons other than wAMD (such as diabetic retinopathy, pathological myopia, retinal vein occlusion, angioid streak disease, ocular histoplasmosis, trauma, etc.), and a history of macular pathology unrelated to wAMD;
4. Any intraocular surgery is planned for the study eye during the study period;
5. The study eye currently has retinal angiomatous proliferation (RAP), central serous chorioretinopathy or symptomatic vitreomacular traction syndrome;
6. Presence of glaucoma or optic neuropathy that involves or compromises the central visual field of the study eye or presence of uncontrolled high intraocular pressure in the study eye；
7. The fellow eye meets the definition of legal blindness；
8. Hormone-induced increased intraocular pressure in any eye；
9. Active infection in any eye this trial (such as those who cannot understand and comply with the trial requirements or are deemed unsuitable for safety reasons).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-16 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability after EXG202 injection | Up to 52 weeks after treatment
  Type, severity, and incidence of adverse events (AEs) and serious adverse events (SAEs) from Week 0 to 52, and dose limited toxicity
Preliminary Efficancy after EXG202 injection | Up to 52 weeks after treatment
  The Best Corrected Visual Acuity (BCVA) change from baseline

SECONDARY OUTCOMES:
Safety and tolerability after EXG202 injection | Up to 24 weeks after treatment
  Type, severity, and incidence of adverse events (AEs) and serious adverse events (SAEs) from Week 0 to 24, and dose limited toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Mingwei ZHAO, PhD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No